CLINICAL TRIAL: NCT07313436
Title: VitaKey Extended Release Protein Dosing
Brief Title: Extended Release Protein Dosing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VitaKey Inc. (Industry)
Collaborators: United States Department of Defense (DOD) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: CLP0001
Record Dates: First submitted 2025-12-03; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Nutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator)
  Interventions: Other: Control
- Low Dose Extended Release Protein (Experimental)
  Interventions: Other: Extended release nutritional protein
- High Dose Extended Release Protein (Experimental)
  Interventions: Other: Extended release nutritional protein
- Negative Dose Extended Release Protein (Experimental)
  Interventions: Other: Negative Dose

INTERVENTIONS:
Other: Extended release nutritional protein — Participants will consume a beverage with extended release protein.
  Arms: High Dose Extended Release Protein; Low Dose Extended Release Protein
Other: Control — Participants will consume a beverage with standard nutritional protein.
  Arms: Control
Other: Negative Dose — Participants will consume a beverage with 15g less extended release protein than either the low dose cohort or the high dose cohort.
  Arms: Negative Dose Extended Release Protein

SUMMARY:
The overall goal of this study is to determine the minimum dose required to elicit measurable elevation of plasma essential amino acid levels 12 hours after consuming VitaKey's extended release protein technology. The results of this study will be used to set a dose for future protein clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 - 40 years of age, inclusive.
2. Body mass index (BMI) of 20 - 28 kg/m2, inclusive.
3. Non-user of tobacco or nicotine products (e.g., cigarette smoking, vaping, chewing tobacco) within 12 months of Visit 1, with no plans to begin use during the study period.
4. Score of 7 to 10 on the Vein Access Scale at Visit 1.
5. No health conditions that would prevent him/her from fulfilling the study requirements as judged by the Clinical Investigator on the basis of medical history.
6. Willing to adhere to all study procedures, including lifestyle considerations (see section 6.3), and sign forms providing informed consent to participate in the study and authorization to release relevant protected health information to the Clinical Investigator.

Exclusion Criteria:

General health related criteria

1. Currently in a habitual exercise training program (≥ 3 d/wk of structured exercise) or plans to initiate an exercise training program during the study period.
2. Uncontrolled hypertension (systolic blood pressure ≥140 mm Hg or diastolic blood pressure ≥90 mm Hg) as defined by the blood pressure measured at visit 1. Stable use of hypertension medication is allowed (defined as no change in medication regimen ≤ 90 d of visit 1).
3. History or presence of clinically important cardiac, renal, hepatic, endocrine, pulmonary, biliary, pancreatic, or neurological disorders that may affect the participant's ability to adhere to the study protocol and/or affect study outcomes, in the judgment of the Investigator.
4. Female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
5. Any signs or symptoms of active infection of clinical relevance (e.g., urinary tract or respiratory) within 5 days prior to any test visit. If an infection occurs during the study period, test visits should be rescheduled until all signs and symptoms have resolved and any treatment has been completed at least 5 d prior to testing.
6. History or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
7. History of any major trauma or major surgical event within 2 months of visit 1.
8. History of an eating disorder (e.g., anorexia nervosa, bulimia nervosa, or binge eating) diagnosed by a health professional.

   Exclusionary products related criteria
9. Recent history of (within 12 months of screening; visit 1) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
10. Recent use of anti-hyperglycemic (e.g., metformin, insulin, DPP 4 inhibitors, SGLT-2 inhibitors, GIP agonist, Pioglitazone, or Sulfonylureas) or GLP-1 analogue (e.g., Ozempic or Wegovy semaglutide, Mounjaro trizapatide) prescription medications within 6 mo of visit 1.
11. Unstable use of any prescription medication, where stable use is defined as no change in dose or medication type within 90 d of visit 1.
12. Exposed to any non-registered drug product within 30 d of visit 1.
13. Antibiotic use within 30 d of visit 1 and throughout the study period.
14. Steroid use within 30 d of visit 1 and throughout the study period.
15. Current habitual user (≥ 3 days/week ≤ 30 d of visit 1) of anti-inflammatory medications (e.g., NSAIDs, acetaminophen, etc.).
16. Habitual users (i.e., daily or almost daily) of marijuana and hemp products, including CBD products. Occasional use (e.g., couple times a month) within 12 months of visit 1 is allowed but requires at least a 14 d washout prior to visit 1 and the participant must be willing to refrain from use during the study (sleep aids and topical lotions/creams are allowed).

    General safety related criteria
17. Known allergy or sensitivity to any ingredients or potential allergens contained in the study product or standard meals.
18. Self-report of blood donation totaling between 101-449 mL of blood within 30 d prior to visit 1 or a blood donation of ≥450 mL within 56 days prior to visit 1, or plasma donations within 48 h of visit 1. As well as any plans to donate blood or plasma during the study period.
19. Any condition the Investigator believes would interfere with the participant's ability to provide informed consent or comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Plasma EAA positive incremental AUC5-12h (calculated as AUC0-12h - AUC0-5h) 5-12 h post-product consumption | 5-12 hours post consumption

SECONDARY OUTCOMES:
Percent change in plasma leucine concentrations | pre-product (t = 0) to 5 hours post consumption
Positive incremental AUC0-12h 0-12 h post-product consumption and individual serum levels of Amylin. | 0-12 hours post consumption
Maximum postprandial baseline-adjusted GI VAS scores over the 12 h in-clinic period (Overall abdominal symptoms, Abdominal bloating, Abdominal pain, Flatulence, Burping, Stomach rumbling, Nausea, Fatigue) | 0-12 hours post consumption
Positive incremental AUC6-12h composite {[desire to eat + hunger + (100 - fullness) + prospective consumption]/4} appetite scores | 6-12 hours post consumption
Positive incremental AUC6-12h food craving scores 6-12 h post-product: (Satisfaction, Thirst, Desire to snack, Food cravings, Sweet cravings, Salty cravings, Savory cravings, Fatty cravings) | 6 - 12 hours post consumption
48 h GI VAS scores [0 to 100 with 0 indicating no symptoms], representing the time since leaving the clinic | 48 hours post consumption
Positive incremental AUC0-12h 0-12 h post-product consumption and individual serum levels of Ghrelin. | 0-12 hours post consumption
Positive incremental AUC0-12h 0-12 h post-product consumption and individual serum levels of GIP. | 0-12 hours post consumption
Positive incremental AUC0-12h 0-12 h post-product consumption and individual serum levels of GLP-1. | 0-12 hours post consumption
Positive incremental AUC0-12h 0-12 h post-product consumption and individual serum levels of Glucagon. | 0-12 hours post consumption
Positive incremental AUC0-12h 0-12 h post-product consumption and individual serum levels of IL-6. | 0-12 hours post consumption
Positive incremental AUC0-12h 0-12 h post-product consumption and individual serum levels of Insulin. | 0-12 hours post consumption
Positive incremental AUC0-12h 0-12 h post-product consumption and individual serum levels of Leptin. | 0-12 hours post consumptio
Positive incremental AUC0-12h 0-12 h post-product consumption and individual serum levels of MCP-1. | 0-12 hours post consumption
Positive incremental AUC0-12h 0-12 h post-product consumption and individual serum levels of PP. | 0-12 hours post consumption
Positive incremental AUC0-12h 0-12 h post-product consumption and individual serum levels of PYY. | 0-12 hours post consumption
Positive incremental AUC0-12h 0-12 h post-product consumption and individual serum levels of TNFα | 0-12 hours post consumption
Individual Hunger appetite scores 6-12 h post-product | 6-12 hours post consumption
Desire to eat individual appetite scores 6-12 h post-product | 6-12 hours post consumption
Fullness individual appetite scores 6-12 h post-product. | 6-12 hours post consumption
Fullness individual appetite scores 6-12 h post-product | 6-12 hours post consumption
Prospective food consumption individual appetite scores 6-12 h post-product | 6-12 hours post consumption

CONTACTS AND LOCATIONS:
Locations (1):
- Biofortis, Addison, Illinois, United States